CLINICAL TRIAL: NCT03586596
Title: Decídetext: Mobile Cessation Support for Latino Smokers
Brief Title: Mobile Cessation Support for Latino Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Lombardi Comprehensive Cancer Center (Other); Children's Mercy Hospital Kansas City (Other); University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Paula Cupertino, Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro2017-0528
Record Dates: First submitted 2018-07-02; First posted 2018-07-13 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Smoking Cessation
Keywords: Smokers; Mobile intervention; Latino; Promotores de Salud; Pharmacotherapy; Cultural accomodation; Tobacco use; Health Disparities; Cancer Disparities
MeSH Terms: conditions — Smoking Cessation; Tobacco Use

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Decídetext program (Experimental): Participants will receive a tablet-based interactive educational session, 6 months of text-messaging based counseling, which includes prompts to access free pharmacotherapy.
  Interventions: Behavioral: The Decídetext program
- Standard Care Control (Active Comparator): Participants will receive an adapted version of standard printed smoking cessation educational materials from the American Cancer Society and, the National Cancer Institute, which include information about the health risks of smoking, benefits & strategies for quitting and access to free pharmacotherapy by calling a free number.
  Interventions: Behavioral: Standard Care Control

INTERVENTIONS:
Behavioral: The Decídetext program — Decídetext participants will be directed to the tablet-based software. Participants will receive an interactive education session that will lead them through language-appropriate, culturally-relevant information about stopping smoking, collection of basic smoking history data, and choices/plans about preparing to quit. Quit plans include: 1) choice of quit date, 2) NRT preference, 3) plan to remove smoking cues, 4) identification of trigger situations and 5) choice of suggested coping strategies. Participant data and choices are used to generate a printed 1-page individualized treatment plan. Tablet components, assessment items, audio narrative, brief multimedia instructional video clips, and the printed treatment plan have been developed to address low-literacy levels.
  Arms: The Decídetext program
Behavioral: Standard Care Control — Educational Material provided as of suggested by American Cancer Society and, the National Cancer Institute
  Arms: Standard Care Control

SUMMARY:
The primary aim of this study is to examine the efficacy of Decídetexto, an innovative mobile smoking cessation intervention that incorporates two elements: 1) a tablet-based e-Health platform that collects personal smoking-related information to support the development of an individualized quit plan and guides the ensuing text messaging program; and 2) a 12-week text messaging "skills-based counseling" (I.e, behavioral support) program that includes educational information, behavioral strategies, motivational messaging, and pharmacotherapy support driven by information obtained from both the tablet program and the user's text messages. The investigators will evaluate its efficacy relative to a standard care condition that provides high quality printed smoking cessation materials along with referral to telephone quit line counseling. Participants in both groups are given access to free pharmacotherapy via a toll-free study number. Experienced Promotores de Salud (Community Health Workers) will use community and clinic-based outreach to recruit Latino smokers into the study. Participants in both conditions will complete follow-up assessment at the end of treatment (Week 12) and Month 6 (primary outcome). Our hypothesis is that at month 6, smokers in Decídetexto will have significantly higher cotinine-verified 7-day point prevalence abstinence (no cigarettes in the past 7 days) than smokers in the control arm.

DETAILED DESCRIPTION:
Latinos are less likely than non-Hispanic whites to have access to healthcare, to have knowledge of existing smoking cessation resources, to receive advice to stop smoking, and to utilize pharmacotherapy to stop smoking. Despite these marked tobacco-related disparities, there is a lack of effective interventions designed for the Latino community. Mobile technology provides a promising method for overcoming barriers and providing culturally congruent treatment to Latino smokers. Implementation of mobile interventions among Latinos remains minimal despite the fact that Latinos are the fastest adopters of mobile technology, utilizing smartphones and text messaging at a higher rate than non-Hispanic whites do. An effective, culturally appropriate intervention using mobile technologies methods with the potential for widespread adoption by clinic and community-based service providers could dramatically increase reach and impact on Latino health.

Decídetext is a culturally congruent method for increasing access to cessation services for Latino smokers and helping them develop, implement, and follow a personalized quit plan. If successful, this intervention could be readily implemented in different settings including community settings, clinics, pharmacies, emergency rooms, and clinic waiting areas and reduce treatment disparities, reduce tobacco-related morbidity and mortality, and improve the health and quality of life for approximately 9 million of Latino smokers in the United States.

Aim 1. To evaluate the impact of the culturally accommodated Decídetext program versus standard care on smoking abstinence at Month 6 among Latino smokers. At Month 6, smokers in Decídetext will have significantly higher cotinine-verified 7-day point prevalence abstinence (no cigarettes in the past 7 days) than smokers in the control arm. Program efficacy also will be examined at Week 12 (end of treatment) to assess mechanisms of change, and Month 12 to provide extended outcome data.

Aim 2. To assess therapeutic alliance, pharmacotherapy utilization, and self-efficacy as mediators of the presumed treatment effect on cotinine-verified 7-day smoking abstinence at Month 6 among Latino smokers. Our hypothesis is that Decídetext will have greater efficacy for smoking cessation than standard care by increasing therapeutic alliance, utilization of pharmacotherapy, and self-efficacy to quit.

Aim 3. To conduct a process evaluation that can inform findings and future improvements. The evaluation of Decídetext includes: 1) satisfaction with the program and its components; 2) text-message system utilization patterns and common content themes in text message interactions among participants.

ELIGIBILITY:
Inclusion Criteria:

* Are you Hispanic or Latino?
* Do you know how to read and speak English and/or Spanish?
* Are you at least 21 years old?
* Have you smoked cigarettes for at least 6 months?
* Within a typical week, how many days do you smoke (even a puff)?
* Within a typical week, how many days do use other tobacco products?
* Are you interested in quitting smoking in the next 30 days?
* Are you currently participating in any other smoking cessation program or taking any type of medication to quit smoking?
* Is any household member participating in this study?
* Are you pregnant, breast-feeding or planning to become pregnant in the next year?
* Are you planning to move out of your current address in the following six months?
* Do you have an active cellphone with unlimited text messaging capability?
* Are you willing to come to 2 study visit, at the beginning and 6 month, and get at least 1 phone calls between visits?
* Do you know how to send/read text messages?
* Is the participant ELIGIBLE? If NOT ELIGIBLE, complete demographics If ELIGIBLE, complete contact information.

Exclusion Criteria:

* Include plans to move from New Jersey in the next 6 months
* If another household member enrolled in the study.
* If answers no to any question of the Eligibility form.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 457 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2021-09-08 (Actual); Study Completion 2021-09-08 (Actual)

PRIMARY OUTCOMES:
Cotinine-verified 7-day point prevalence at 6 months. | 6 months
  Participants who quit will do a cotinine-verified 7-day point prevalence check at Month 6.

SECONDARY OUTCOMES:
12- week self-report | 12 weeks
  Participants in both conditions will complete follow-up assessment at the end of the treatment at 12 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Paula Cupertino, PhD, Principal Investigator — University of Rochester
Locations (3):
- United States (3):
  - University of Kansas Medical Center, Kansas City, Kansas
  - Hackensack Meridian Health - Hackensack University Medical Center, Hackensack, New Jersey
  - University of Rochester Medical Center, Rochester, New York

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] 1. Blanco L, Garcia R, Perez-Stable E, et al. National trends in smoking behaviors among Mexican, Puerto Rican, and Cuban men and women in the United States. American Journal of Public Health. 2014;104(5):896-903. 2. CDC. Cigarette smoking among adults and trends in smoking cessation - United States, 2008. Morbidity and Mortality Weekly Report (MMWR) 2009;58(44):1227-1232. 3. Trinidad D, Pérez-Stable E, White M, Emery S, Messer K. A nationwide analysis of US racial/ethnic disparities in smoking behaviors, smoking cessation, and cessation-related factors. American Journal of Public Health. 2011;101(4):699-706. 4. Duggan M. Cell Phone Activities 2013. Pew Research Center; September 2013 2013. 5. Anderson M. Technology device ownership: 2015. Pew Research Center; October, 2015 2015. 6. Burrow-Sanchez JJ, Martinez CR, Hops H, Wrona M. Cultural accommodation of substance abuse treatment for Latino adolescents. Journal of Ethnicity in substance abuse. 2011;10(3):202-225.
- [Background] 7. Colby S, Ortman J. Projections of the Size and Composition of the U.S. Population: 2014 to 2060: Population Estimates and Projections. 2015. 8. Bethel JW, Schenker MB. Acculturation and smoking patterns among Hispanics: a review. American Journal of Preventive Medicine. 2005;29(2):143-148. 9. Lee D, Fleming L, Arheart K, et al. Smoking rate trends in U.S. occupational groups: The 1987 to 2004 National Health Interview Survey. Journal of Occupational and Environmental Medicine. 2007;49(1):75-81. 10. Wilkinson AV, Spitz MR, Strom SS, et al. Effects of nativity, age at migration, and acculturation on smoking among adult Houston residents of Mexican descent. American Journal of Public Health. 2005;95(6):1043-1049. 11. CDC. CDC Health disparities and inequalities report - United States, 2011. Morbidity and Mortality Weekly Report (MMWR). 2011;60:109-113.
- [Background] 12. CDC. Targeting tobacco use: the nation's leading cause of death 2004. Atlanta: United States Department of Health and Human Services;2004. 13. Shalala D, Broome C, Satcher D. Tobacco Use Among U.S. Racial/Ethnic Minority Groups - African Americans, American Indians and Alaska Natives, Asian Americans, Pacific Islander and Hispanics: A report of the Surgeon General. 1998. 14. Smith BD, Smith GL, Hurria A, Hortobagyi GN, Buchholz TA. Future of cancer incidence in the United States: burdens upon an aging, changing nation. Journal of Clinical Oncology. 2009;27(17):2758-2765. 15. Webb MS, Rodríguez-Esquivel D, Baker EA. Smoking cessation interventions among Hispanics in the United States: A systematic review and mini meta-analysis. American Journal of Health Promotion. 2010;25(2):109-118. 16. Lewin ME, Baxter RJ. America's health care safety net: revisiting the 2000 IOM report. Health affairs (Project Hope). 2007;26(5):1490-1494.
- [Background] 17. Maher JE, Rohde K, Dent CW, et al. Is a statewide tobacco quitline an appropriate service for specific populations? Tobacco Control. 2007;16 Suppl 1:i65-70. 18. Zuniga E, Castaneda, X., Averbach, A., & Wallace, S.P. Mexican and Central American immigrants in the United State: Health care access. . Regents of the University of California and the Mexican Secretariat of Health. 2006. 19. CDC. Quitting Smoking Among Adults - United States, 2001 - 2010. Atlanta, GA: Center for Disease Control and Prevention;2011. 20. Soto Mas FG, Papenfuss RL, Jacobson HE, Hsu CE, Urrutia-Rojas X, Kane WM. Hispanic physicians' tobacco intervention practices: a cross-sectional survey study. BMC Public Health. 2005;5:120. 21. Zhu K, Levine RS, Brann EA, Gnepp DR, Baum MK. A population-based case-control study of the relationship between cigarette smoking and nasopharyngeal cancer (United States). Cancer Causes Control. 1995;6(6):507-512.
- [Background] Sherrill W, Crew L, Mayo RB, Mayo WF, Rogers BL, Haynes DF. Educational and health services innovation to improve care for rural Hispanic communities in the USA. Rural Remote Health. 2005 Oct-Dec;5(4):402. Epub 2005 Nov 11. PMID 16283825
- [Background] 26. Foraker RE, Patten CA, Lopez KN, Croghan IT, Thomas JL. Beliefs and attitudes regarding smoking among young adult Latinos: a pilot study. Preventive Medicine. 2005;41(1):126-133. 27. Team. DREGaNDP. Tobacco use in Minnesota: perspectives from Latino communities. Executive summary. Minnesota. : Blue Cross and Blue Shield of Minnesota, Communidades Latinas Unidas en Servicio, Minnesota Partnership for Action Against Tobacco;2006. 28. Bock BC, Niaura RS, Neighbors CJ, Carmona-Barros R, Azam M. Differences between Latino and non-Latino White smokers in cognitive and behavioral characteristics relevant to smoking cessation. Addictive Behaviors. 2005;30(4):711-724. 29. Fiore M, Jaen, CR, Baker, TB. Treating tobacco use and dependence: 2008 update. Rockville, MD: U.S. Department of Health and Human Services; 2008. 30. Cox L, Okuyemi K, Choi W, Ahluwalia J. A review of tobacco use treatments in U.S. ethnic minority populations. American Journal of Health Promotion. 2011;25(5S):S11-S30.
- [Background] 31. Webb M, Rogers BG, Okuyemi K. Smoking cessation among racial/ethnic minorities, 2010-2014. Current Addiction Reports. 2015;2(1):24-32. 32. Leischow SJ, Hill A, Cook G. The effects of transdermal nicotine for the treatment of Hispanic smokers. American Journal of Health Behavior. 1996;20(5):304-311. 33. Woodruff SI, Talavera GA, Elder JP. Evaluation of a culturally appropriate smoking cessation intervention for Latinos. Tobacco Control. 2002;11(4):361-367. 34. Kreps GL, Neuhauser L. New directions in eHealth communication: opportunities and challenges. Patient education and counseling. 2010;78(3):329-336. 35. Cole-Lewis H, Kershaw T. Text messaging as a tool for behavior change in disease prevention and management. Epidemiologic Reviews. 2010;32:56-69. 36. Whittaker R, McRobbie H, Bullen C, Borland R, Rodgers A, Gu Y. Mobile phone-based interventions for smoking cessation. The Cochrane database of systematic reviews. 2012;11.
- [Background] 37. Heron KE, Smyth JM. Ecological momentary interventions: incorporating mobile technology into psychosocial and health behaviour treatments. British journal of health psychology. 2010;15(1):1-39. 38. Kim BH, Glanz K. Text messaging to motivate walking in older African Americans: a randomized controlled trial. American Journal of Preventative Medicine. 2013;44(1):71-75. 39. Gerber BS, Stolley MR, Thompson AL, Sharp LK, Fitzgibbon ML. Mobile phone text messaging to promote healthy behaviors and weight loss maintenance: a feasibility study. Health Informatics Journal. 2009;15(1):17-25. 40. Patrick K, Raab F, Adams MA, et al. A text message-based intervention for weight loss: randomized controlled trial. Journal of Medical Internet Research. 2009;11(1):e1. 41. Rodgers A, Corbett T, Bramley D, et al. Do u smoke after txt? Results of a randomised trial of smoking cessation using mobile phone text messaging. Tobacco Control. 2005;14(4):255-261.
- [Background] Naditz A. Medication compliance--helping patients through technology: modern "smart" pillboxes keep memory-short patients on their medical regimen. Telemed J E Health. 2008 Nov;14(9):875-80. doi: 10.1089/tmj.2008.8476. No abstract available. PMID 19062349
- [Background] 43. Krishna S, Boren SA. Diabetes self-management care via cell phone: a systematic review. Journal of diabetes science and technology. 2008;2(3):509-517. 44. Free C, Phillips G, Watson L, et al. The effectiveness of mobile-health technologies to improve health care service delivery processes: a systematic review and meta-analysis. PLOs Medicine. 2013;10(1):e1001362. 45. Kong G, Ells D, Camenga D, Krishnan-Sarin S. Text messaging-based smoking cessation intervention: A narrative review. Addictive Behaviors. 2014;39(5):907-917. 46. De Leon E, Fuentes L, Cohen J. Characterizing periodic messaging interventions across health behaviors and media: systematic review. Journal of Medical Internet Research. 2014;16(3):e93. 47. Brendryen H, Drozd F, Kraft P. A digital smoking cessation program delivered through internet and cell phone without nicotine replacement (happy ending): randomized controlled trial. Journal of Medical Internet Research. 2008;10(5):e51.
- [Background] 48. Abroms L, Boal A, Simmens S, Mendel J, Windsor R. A randomized trial of Text2Quit: a text messaging program for smoking cessation. American Journal of Preventative Medicine. 2014;47(3):242-250. 49. Fox S, Livingston G. Latinos Online: Hispanics with lower level of education and English proficiency remain largely disconnected from the Internet. Washington, DC: Pew Internet and American Life Project & Pew Hispanic Center;2007. 50. Zickuhr K. Generations 2010. Washington, D.C.2010. 51. Tarnowski J. Opiniones 2007: Hispanics respond well to direct mail, text messaging. Vertis Communication 2007. 52. Ahlers-Schmidt CR, Ablah E, Rogers N, et al. Low-Income Urban Latino Parents' Perceptions of Immunization Text Reminders. Ethnicity and Disease. 2013:229-235. 53. Group TTRI. Tobacco research implementation plan. Priorities for tobacco research beyond the year 2000. . Bethesda, MD: National Cancer Institute, National Institute of Health.;1998.
- [Background] Free C, Phillips G, Galli L, Watson L, Felix L, Edwards P, Patel V, Haines A. The effectiveness of mobile-health technology-based health behaviour change or disease management interventions for health care consumers: a systematic review. PLoS Med. 2013;10(1):e1001362. doi: 10.1371/journal.pmed.1001362. Epub 2013 Jan 15. PMID 23349621
- [Background] 60. Bordin ES. Theory and research on the therapeutic working alliance: New directions. The working alliance: Theory, research, and practice. 1994:13-37. 61. Ardito RB, Rabellino D. Therapeutic alliance and outcome of psychotherapy: Historical excursus, measurements, and prospects for research. Frontiers in psychology. 2011;2(1):270. 62. Horvath AO, Symonds BD. Relation between working alliance and outcome in psychotherapy: A meta-analysis. Journal of counseling psychology. 1991;38(2):139. 63. Cupertino AP, Berg C, Azor Hui SK, Richter K, Gajewski BJ, Ellerbeck EF. Change in Self-Efficacy, Autonomous and Controlled Motivation Predicting Smoking Cessation. Society for Research on Nicotine and Tobacco; 2010; Baltimore, MD.
- [Background] 64. Suarez N, Cox L, Richter K, et al. Success of "Promotores de Salud" in identifying immigrant Latino smokers and developing quit plans In: Caron R, Merrick J, eds. Building Community Capacity: Minority and Immigrant Populations. Hauppauge, New York: Nova Science Publishers 2012:343. 65. Cupertino AP, Fernandez C, Reynoso E, et al. Reinforcing promotores de salud and a culturally appropriate quit smoking program. Promotores de Salud Annual Conference; 2010; San Francisco, CA. 66. Fernandez C, Bullard E, Cupertino AP, Morgan A, Mendoza I, Garrett S. Promotores de salud: community-based model to address health disparities among Latinos. KDHE Center for Health Disparities Conference.; 2009; Topeka, KS. 67. Saint-Elin M, Bravo J, Estrella O, et al. Promotores de salud program in Southwest Kansas. Kansas City, KS: Juntos Center for Advancing Latino Health February 2012.
- [Background] 68. Sechrest L. Opening access to tobacco dependence treatment resources for Spanish-speaking cessation providers in the U.S. Mexico border region: promotores contra el tabaco en la frontera. Tucson, Arizona: The University of Arizona;2006. 69. Cupertino AP, Wick JA, Richter KP, Mussulman L, Nazir N, Ellerbeck EF. The impact of repeated cycles of pharmacotherapy on smoking cessation: a longitudinal cohort study. Archives of Internal Medicine. 2009;169(20):1928-1930. PMCID: 2826277 70. Cupertino AP, Richter K, Cox LS, et al. Feasibility of a Spanish / English computerized decision aid to facilitate smoking cessation efforts in underserved communities. Journal of Health Care for the Poor and Underserved 2010;21:504-517. PMID: 20453353 71. Engelman KK, Cupertino AP, Daley CM, et al. Engaging diverse underserved communities to bridge the mamography divide. Public Health. 2011;11:47. PMCID: 3036625.
- [Background] 72. Cox LS, Wick JA, Nazir N, et al. Predictors of early versus late smoking abstinence within a 24-month disease management program. Nicotine and Tobacco Research. 2011;13(3):215-220. 73. Cox LS, Cupertino AP, Tercyak KP. Interest in participating in smoking cessation programs among Latino primary care patients. Journal of Clinical Psychology in Medical Settings 2011. PMCID: 3229918 74. Cupertino AP, Richter KP, Cox LS, et al. Smoking cessation pharmacotherapy preferences in rural primary care. Nicotine and Tobacco Research. 2008;10(2):301-307. PMCID: 2821185 75. Sheppard VB, Cox LS, Kanamori MJ, et al. Brief report: if you build it, they will come: methods for recruiting Latinos into cancer research. Journal of General Internal Medince. 2005;20(5):444-447.
- [Background] 76. Cox LS, Feng S, Canar J, McGlinchey Ford M, Tercyak KP. Social and behavioral correlates of cigarette smoking among mid-Atlantic Latino primary care patients. Cancer Epidemiology, Biomarkers and Prevention. 2005;14(8):1976-1980. 77. Cox LS, Nollen N, Mayo MS, et al. Bupropion for Smoking Cessation in African American Light Smokers: A Randomized Controlled Trial. Journal of the National Cancer Institute. 2012;104:1-9. 78. Champassak SL, Goggin K, Finocchario-Kessler S, et al. A qualitative assessment of provider perspectives on smoking cessation counselling. Journal of evaluation in clinical practice. 2014;20(3):281-287. 79. Choi WS, Faseru B, Beebe LA, et al. Culturally-tailored smoking cessation for American Indians: study protocol for a randomized controlled trial. Trials. 2011;12(1):126.
- [Background] 80. Wearing J, Nollen N, Befort C, Davis A, Agemy C. iPhone app adherence to expert-recommended guidelines for pediatric obesity prevention. Childhood Obesity. 2014;10(2):132-144. 81. Ellerbeck EF, Mahnken JD, Cupertino AP, et al. Effect of varying levels of disease management on smoking cessation: a randomized trial. Annals of Internal Medicine. 2009;150(7):437-446. 82. Cupertino AP, Suarez N, Cox LS, et al. Empowering Promotores de Salud to engage in Community-Based Participatory Research Journal of Immigrant and Refugee Studies. 2013;11(1):24-43. PMCID: 4335649 83. Cupertino AP, Cox LS, Garrett S, et al. Tobacco Use and Interest in Smoking Cessation among Latinos Attending Community Health Fairs. Journal of Immigrant and Minority Health. 2010;13(4):719-724.
- [Background] 84. Cupertino AP, Saint-Elin M, Bravo de los Rios J, Greiner A. Empowering promotores de salud as partners in advancing knowledge and participation in cancer research studies. American Association for Cancer Research; 2013; San Diego, CA. 85. Luoto R, Uutela A, Puska P. Occasional smoking increase total and cardiovascular mortality among men. Nicotine and Tobacco Research. 2000;2(2):133-139. 86. Hayes RB, Borrelli B. Differences between Latino daily light and heavier smokers in smoking attitudes, risk perceptions, and smoking cessation outcome. Nicotine and Tobacco Research. 2013;15(1):103-111. 87. Ayanian JZ, Cleary PD. Perceived risks of heart disease and cancer among cigarette smokers. JAMA. 1999;281(11):1019-1021.
- [Background] 88. Zinzer M, Pampel F, Flores E. Distinct beliefs, attitudes, and experiences of Latino smokers: Relevance for cessation interventions. American Journal of Health Promotion. 2011;25(5S):S1-S15. 89. Tong EK, Ong MK, Vittinghoff E, Perez-Stable EJ. Nondaily smokers should be asked and advised to quit. American Journal of Preventive Medicine. 2006;30(1):23-30. 90. Schane RE, Ling PM, Glantz SA. Health effects of light and intermittent smoking: a review. Circulation. 2010;121(13):1518-1522. 91. Shiffman S, Tindle H, Li X, Scholl S, Dunbar M, Mitchell-Miland C. Characteristics and smoking patterns of intermittent smokers. Experimental and clinical psychopharmacology. 2012;20(4):264. 92. Schauer GL, Malarcher AM, Berg CJ. Differences in smoking and cessation characteristics among adult nondaily smokers in the United States: findings from the 2009-2010 National Adult Tobacco Survey. Nicotine & tobacco research. 2014;16(1):58-68.
- [Background] 93. Reitzel LR, Costello TJ, Mazas CA, et al. Low-level smoking among Spanish-speaking Latino smokers: Relationships with demographics, tobacco dependence, withdrawal, and cessation. Nicotine and Tobacco Research. 2009;11(2):178-184. 94. Cupertino AP, Cox LS, Richter K, Ellerbeck EF. A Pilot Study of a Decision-Aid Tool for Smoking Cessation among Latinos. Society of Research Nicotine and Tobacco 2008; Portland, OR. 95. Cox LS, Cupertino AP, Mussulman LM, et al. Design and baseline characteristics from the KAN-QUIT disease management intervention for rural smokers in primary care. Preventive Medicine. 2008;47(2):200-205. PMCID: 2577567 96. Garrett S, Cupertino AP, Cox LS, et al. Tobacco use and interest in smoking cessation among Latinos attending community Health Fairs. Society for Research on Nicotine and Tobacco; 2010; Baltimore, MD.
- [Background] 97. Leon A, Garrett S, Muñoz M, et al. Using Case Management for Smoking Cessation among Latinos. Paper presented at: Society of Research on Nicotine and Tobacco2012; Houston, TX. 98. Pan Y, De la Puente, M. Census Bureau guideline for the translation of data collection instruments and supporting materials. United Stated Bureau of the Census 2005:pp. 38. 99. Harkness JA, Van de Vijver, F.J.R., Mohler, P.P. Questionnaire Translation. Cross-cultural survey research. 2003:pp. 35-56. 100. Hughes JR, Keely JP, Niaura RS, Ossip-Klein DJ, Richmond RL, Swan GE. Measures of abstinence in clinical trials: issues and recommendations. Nicotine and Tobacco Research. 2003;5(1):13-25. 101. Benowitz N, Ahijevych K, Jarvis MJ, et al. Biochemical verification of tobacco use and cessation. Nicotine and Tobacco Research. 2002;4:149-159.
- [Background] 102. Jarvis MJ, Tunstall-Pedoe H, Feyerabend C, Vesey C, Saloojee Y. Comparison of tests used to distinguish smokers from nonsmokers. American Journal of Public Health. 1987;77(11):1435-1438. 103. Abrams DB, Follick MJ, Biener L, Carey KB, Hitti J. Saliva cotinine as a measure of smoking status in field settings. Am J Public Health. 1987;77(7):846-848. 104. Benowitz NL, Bernert JT, Caraballo RS, Holiday DB, Wang J. Optimal serum cotinine levels for distinguishing cigarette smokers and nonsmokers within different racial/ethnic groups in the United States between 1999 and 2004. American Journal of Epidemiology. 2009;169(2):236-248. 105. Nelson D. Reliability and validity of measures from the Behavioral Risk Factor Surveillance System (BRFSS). Sozial und Praventivmedizin 2001;46(1):S3-42.
- [Background] 106. Hymowitz N, Corle D, Royce J, et al. Smokers' baseline characteristics in the COMMIT trial. Preventive Medicine. 1995;24(5):503-508. 107. Lewis-Esquerre JM, Colby SM, Tevyaw TO, Eaton CA, Kahler CW, Monti PM. Validation of the timeline follow-back in the assessment of adolescent smoking. Drug Alcohol Depend. 2005;79(1):33-43. 108. Fagerstrom KO. Measuring degree of physical dependence to tobacco smoking with reference to individualization of treatment. Addictive Behaviors. 1978;3(3-4):235-241. 109. Marín G, Sabogal, F., Marin, B., Otero-Sabogal, R., Pérez-Stable, E.J. . Development of a short acculturation scale for Hispanics. Hispanic Journal of Behavioral Sciences. 1987; 9,:183-205. 110. Tomas-Sabado J, Qureshi A, Antonin M, Collazos F. Construction and preliminary validation of the Barcelona Inmigration Stress Scale Psychological Reports. 2007;100:1013-1023.
- [Background] 111. Velicer WF, DiClemente CC, Rossi JS, Prochaska JO. Relapse situations and self-efficacy: An integrative model. Addictive behaviors. 1990;15(3):271-283. 112. Hatcher RL, Gillaspy JA. Development and validation of a revised short version of the Working Alliance Inventory. Psychotherapy Research. 2006;16(1):12-25. 113. Abroms L, Hershcovitz R, Boal A, Levine H. Feasibility and acceptability of a text messaging program for smoking cessation in Israel. Journal of Health Communication. 2015;20(8):903-909. 114. Munoz RF, Marin BV, Posner SF, Perez-Stable EJ. Mood management mail intervention increases abstinence rates for Spanish-speaking Latino smokers. American Journal of Community Psychology. 1997;25(3):325-343.
- [Background] 115. Nevid JS, Javier RA. Preliminary investigation of a culturally specific smoking cessation intervention for Hispanic smokers. American Journal of Health Promotion. 1997;11(3):198-207. 116. Baron RM, A. KD. The moderator-mediator variable distinction in social psychological research: Conceptual, strategic, and statistical considerations. Journal of Personality and Social Psychology. 1986;51(6):1173-1182. 117. MacKinnon D. Analysis of mediating variables in prevention and intervention research. NIDA Research Monograph. 1994;139:127-153. 118. Muthén LK, Muthén BO. Mplus User's Guide. 7th ed. Los Angeles, CA: Muthén & Muthén; 1998-2012.
- [Background] Diaz FJ, Perez-Iglesias R, Mata I, Martinez-Garcia O, Vazquez-Barquero JL, de Leon J, Crespo-Facorro B. Using structural equations to test for a direct effect of some antipsychotics on triglyceride levels in drug-naive first-episode psychosis patients. Schizophr Res. 2011 Sep;131(1-3):82-9. doi: 10.1016/j.schres.2011.06.006. Epub 2011 Jul 2. PMID 21726981
- [Background] 123. Hu L, Bentler P. Fit indices in covariance structure modeling: Sensitivity to underparameterized model misspecification. Psychological Methods. 1998;3(4):424-453. 124. Steiger J. Structural model equation and modification: An interval estimation approach. Multivariate Behavioral Research. 1990;25(2):173-180. 125. Tucker L, Lewis C. A reliability coefficient for maximum likelihood factor analysis. Psychometrika. 1973;38(1):1-10. 126. StataCorp. Stata Statistical Software: Release 13. College Station, TX2013.
- [Derived] Cartujano-Barrera F, Cox LS, Catley D, Cai X, Diaz FJ, Arana-Chicas E, Chavez-Iniguez A, Ogedegbe C, Graves KD, Rivera MP, Ponce A, Ellerbeck EF, Cupertino AP. Decidetexto: Mobile Cessation Support for Latino Adults Who Smoke: A Randomized Clinical Trial. Chest. 2025 Feb;167(2):619-629. doi: 10.1016/j.chest.2024.07.160. Epub 2024 Aug 10. PMID 39134144
- [Derived] Arana-Chicas E, Cartujano-Barrera F, Rieth KK, Richter KK, Ellerbeck EF, Cox LS, Graves KD, Diaz FJ, Catley D, Cupertino AP. Effectiveness of Recruitment Strategies of Latino Smokers: Secondary Analysis of a Mobile Health Smoking Cessation Randomized Clinical Trial. J Med Internet Res. 2022 Jun 27;24(6):e34863. doi: 10.2196/34863. PMID 35759320